CLINICAL TRIAL: NCT03399513
Title: Ibrutinib and Standard Immuno-Chemotherapy (R-CHOEP-14) in Younger, High-Risk Patients With Diffuse Large B-Cell Lymphoma
Brief Title: Ibrutinib and Standard Immuno-Chemotherapy in Younger, High-Risk Patients With Diffuse Large B-Cell Lymphoma
Acronym: R-CHOEP-brut
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM17_0017
Record Dates: First submitted 2017-12-18; First posted 2018-01-16 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Ibrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibrutinib and R-CHOEP chemotherapy (Experimental): All patients will receive 8 cycles of R-CHOEP immunochemotherapy every two weeks with the following doses per cycle: rituximab 375 mg/m², cyclophosphamide 750 mg/m², doxorubicin 50 mg/m², vincristine 1.4 mg/m² (dose capped at 2 mg), etoposide 300 mg/m², prednisolone 500 mg.
  In addition, ibrutinib capsules will be administered orally once daily at a dose of 560 mg (4 x 140 mg hard capsules) for 112 days.
  Interventions: Drug: Ibrutinib Oral Capsule [Imbruvica]; Drug: R-CHOEP chemotherapy

INTERVENTIONS:
Drug: Ibrutinib Oral Capsule [Imbruvica] — Imbruvica 140 mg hard capsules (Active substance: Ibrutinib)
Drug: R-CHOEP chemotherapy — Immunochemotherapy

SUMMARY:
This study will investigate if treatment results obtained with R-CHOEP in young high-risk patients with diffuse large B-cell lymphoma can be further improved by the addition of ibrutinib to this regimen.

DETAILED DESCRIPTION:
Encouraging results have been achieved in younger high-risk patients with newly diagnosed diffuse large B-cell lymphoma treated with R-CHOEP. However, more than one fourth of patients still relapse or show primary progressive disease. The outcome of such patients is poor, in particular if first-line therapy contained rituximab. In order to avoid such detrimental situations, we seek to further improve progression-free survival and overall survival by combining R-CHOEP with ibrutinib.

Ibrutinib is a first-in-class, orally administered, potent, small-molecule inhibitor of Bruton's tyrosine kinase, a mediator of critical B-cell signaling pathways implicated in the pathogenesis of B-cell cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.
2. Age between 18-60 years
3. Risk score 2 or 3 according to age-adjusted International Prognostic Index
4. Histology: Primary diagnosis of diffuse large B-cell lymphoma
5. Performance status: ECOG (toxicity and response criteria of the eastern cooperative oncology group) 0-3
6. Stage: all stages according Ann Arbor
7. Absolute neutrophil count: > 1000 cells/microliter (independent of growth factor support)
8. Platelet count ≥ 100.000/mm³ or ≥ 50.000/mm³ if bone marrow involvement independent of transfusion support in either situation.
9. Alanine-aminotransferase and Aspartate-aminotransferase: < 3 x Upper limit of normal value
10. Total Bilirubin: < 1.5 x Upper limit of normal value
11. Serum Creatinine: < 2 x Upper limit of normal value or estimated Glomerular filtration rate (Glomerular filtration rate [Cockcroft-Gault]) ≥ 40 ml/min
12. Women of childbearing potential and men who are sexually active must be practising a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For male subjects, these restrictions apply for 6 months after last dose of study drug. For female subjects, they apply for 12 months after last dose of study drug.
13. Women of childbearing potential must have negative serum or urine beta-human chorionic gonadotropin pregnancy test at screening. Women who are pregnant or breast-feeding are ineligible for this study.
14. Willing/ able to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

1. Vaccinated with live, attenuated vaccines within 4 weeks of inclusion.
2. Major surgery within 4 weeks of inclusion.
3. Any prior lymphoma-directed therapy (except pre-phase treatment).
4. Known central nervous system involvement.
5. Diagnosed or treated for malignancy other than diffuse large B-cell lymphoma, in particular any other (indolent) lymphoma.
6. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional classification.
7. Bone marrow involvement > 25%
8. History of stroke or intracranial hemorrhage within six months of inclusion.
9. Requires anticoagulation with warfarin or equivalent vitamin K antagonist.
10. Known history of human immunodeficiency virus or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection requiring IV antibiotics.
11. Requires treatment with strong CYP3A inhibitors.
12. Use of preparations containing St. John's Wort.
13. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
14. Concurrent treatment with other investigational agent or X-ray therapy.
15. Previous chemo- or radiotherapy for any other malignancy, in particular indolent lymphoma.
16. Any psychological, cognitive, familial, sociological or geographical condition that, in the investigator's opinion, compromises the patient's ability to understand the patient information, to give informed consent or to comply with the study protocol.
17. Participation in another interventional clinical trial during this trial. There may be exceptions at the discretion of the coordinating investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
2-year progression-free survival | From the day of inclusion into the study until one of the following events occurs, whichever is first: disease progression, relapse, death due to any other cause (assessed up to 4 years).
  Length of time that a patient lives without disease progression or relapse.

SECONDARY OUTCOMES:
Overall survival | From the day of inclusion into the study to death due to any cause (assessed up to 4 years).
  The percentage of patients in this study who are still alive.
Event-free survival | From the day of inclusion into the study until one of the following events occurs, whichever comes first: disease progression, start of additional, unplanned anti-tumor therapy, relapse, death due to any other cause (assessed up to 4 years).
  Length of time that a patient remains free of certain events (disease progression, start of additional, unplanned anti-tumor therapy, relapse, death due to any other cause).
Rate of complete remission | From the day of inclusion into the study until date of complete remission (assessed up to 6 months).
  Rate of complete remission measured as number of complete remissions divided by the number of patients included.
Rate of partial remission | From the day of inclusion into the study until date of partial remission (assessed up to 6 months).
  Rate of partial remission measured as number of partial remissions divided by the number of patients included.
Overall response rate | From the day of inclusion into the study until date of complete or partial remission (assessed up to 6 months).
  Overall response rate measured as number of complete and partial remissions divided by the number of patients included.
Progression rate | From the day of inclusion into the study until date of progression during therapy or within 2 months after last treatment course (assessed up to 6 months).
  Progression rate measured as number of progressions divided by the number of patients included.
Relapse rate | From the day of inclusion into the study until date of relapse during therapy or within 2 months after last treatment course (assessed up to 6 months).
  Relapse rate measured as number of relapses divided by the number of patients included.
Duration of response | From documentation of tumor response to disease progression or relapse (assessed up to 6 months).
  The time between the initial response to therapy and subsequent disease progression or relapse.
Adverse events and serious adverse events | The documentation of adverse events, including serious adverse events, starts with first study treatment after patient inclusion and ends 100 days after the last application of ibrutinib or any component of R-CHOEP (whichever is applied last).
  Frequency of adverse events and serious adverse events
Rate of treatment-related deaths | From the start of therapy up to 2 months after the end of therapy.
  The number of deaths during therapy or up to 2 months after the end of therapy divided by the number of patients who started study treatment.
Therapy cycles (number) | From the start of therapy until the end of therapy (assessed up to 4 months).
  Number of therapy cycles
Therapy cycles (duration) | From the start of therapy until the end of therapy (assessed up to 4 months).
  Duration of therapy cycles
Used drugs | From the start of therapy until the end of therapy (assessed up to 4 months).
  Cumulative doses of R-CHOEP (cyclophosphamide, doxorubicin, vincristine, etoposide, rituximab) and ibrutinib.
Outcome according to lymphoma biology | From the start of study until the end of study (assessed up to 4 years).
  Lymphoma tissue from all patients will be characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Norbert Schmitz, MD, Principal Investigator — University Hospital Muenster
Locations (12):
- Germany (12):
  - HELIOS Hospital Berlin-Buch, Berlin
  - Hospital Chemnitz, Chemnitz
  - University Hospital Cologne, Cologne
  - University Hospital Göttingen, Göttingen
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Saarland University Hospital, Homburg
  - Johannes Wesling Hospital Minden, Minden
  - University Hospital Muenster, Münster
  - Rostock University Medical Center, Rostock
  - University Hospital Tuebingen, Tübingen
  - University Hospital Ulm, Ulm